CLINICAL TRIAL: NCT06685237
Title: CoPenhagen Heart Failure With Preserved Ejection Fraction (CPH-HFpEF)
Brief Title: Copenhagen Heart Failure With Preserved Ejection Fraction
Acronym: CPH-HFpEF
Status: Recruiting | Type: Observational
Sponsor: Tor Biering-Sørensen (Other)
Responsible Party: Sponsor-Investigator, Tor Biering-Sørensen, Professor, Herlev and Gentofte Hospital
Organization: Herlev and Gentofte Hospital (Other)
Other Study IDs: CPH-HFpEF; H-24022361 (Other: De Videnskabsetiske Komitéer for Region Hovedstaden (VEK))
Record Dates: First submitted 2024-11-11; First posted 2024-11-12 (Actual); Last update posted 2025-03-05 (Actual); Status verified 2025-03

CONDITIONS: Heart Failure With Preserved Ejection Fraction (HFPEF)
Keywords: Heart failure with preserved ejection fraction; HFpEF; Registry; Screening; Echocardiography; Questionnaire; NT-proBNP

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood samples.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
Heart failure with preserved ejection fraction (HFpEF) has grown to become the dominant form of heart failure (HF) worldwide, in tandem with ageing of the general population and the increasing prevalence of obesity, diabetes mellitus and hypertension. In 2020, > 70% of patients with heart failure had preserved ejection fraction. The incidence and prevalence of HFpEF has been growing by 10% every 10 years relative to HF with reduced ejection fraction (HFrEF). In 2017, the prevalence of HFpEF varied from 1% to 14% based on available data from Europe and USA. HFpEF is associated with high morbidity and mortality, and patients with HFpEF have similarly high hospitalization rates as patients with HFrEF. Hence, HFpEF poses a substantial global health challenge. Despite its prevalence, HFpEF remains undiagnosed and underrecognized, necessitating a comprehensive approach to both identification and management.

Ensuring successful treatment necessitates early identification of HFpEF. Consequently, a targeted screening strategy has been devised for the identification of HFpEF patients. Given the higher prevalence of heart failure (HF) in the elderly population, testing the screening strategy is imperative to customize it to the specific needs of vulnerable patients who may be more inclined to decline participation in the screening program.

DETAILED DESCRIPTION:
The study is a prospective, observational cohort study. Using risk factors for HFpEF, the Danish National Health Registries will be used to identify up to 5000 citizens with at least one risk factor for HFpEF relying on International Classification of Diseases, 10th revision (ICD-10), medication, and biochemistry. The investigators will only recruit patients from the Capital Region of Denmark. Participants will be recruited by sending recruitment letters to a secure electronic mailbox (eBoks) linked to the patients' social security numbers.

The purpose of this study is to evaluate the identification and screening procedures for HFpEF outlined in this protocol. Additionally, the investigators aim to gauge the willingness of identified Danish adults with risk factors for HFpEF to participate in the study and to identify and address any barriers to their involvement. Overall, the investigators expect the results of this study can be used to guide future initiatives aimed at improving the identification and enrollment of patients with HFpEF, particularly among vulnerable populations.

ELIGIBILITY:
Inclusion Criteria:

1. Residence in the Capital Region of Denmark
2. Age ≥ 50 years
3. At least two risk factors for HFpEF defined as any of the following (for age ≥ 60 years, only one):

   * Hypertension
   * Diabetes mellitus
   * Chronic kidney disease
   * Atrial fibrillation
   * BMI > 25 kg/m2
   * Previous heart valve surgery
   * Ischemic heart disease
   * Obstructive sleep apnea
   * Furosemide 40 mg

Exclusion Criteria:

1. Age ≥ 90 years
2. Prevalent HF
3. Dementia
4. Nursing home
5. Amyloidosis
6. Hemodialysis
7. Cancer diagnosed within the past 5 years (skin cancer not included)
8. Prior solid organ transplantation
9. Lung disease defined as any of the following:

   * World Health Organization Group 1 pulmonary hypertension
   * Chronic pulmonary embolism
   * Lung fibrosis
   * Chronic obstructive pulmonary disease (COPD)
   * Home oxygen

Ages: 50 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 5000 citizens aged 50 years or above in the Capital Region of Denmark with at least two risk factors for HFpEF (for age ≥ 60 years, only one).
Sampling Method: Non-Probability Sample
Enrollment: 5000 (Estimated)
Dates: Start 2025-02-28 (Actual); Primary Completion 2025-11-28 (Estimated); Study Completion 2026-03-28 (Estimated)

PRIMARY OUTCOMES:
The primary objective of this study is to pilot the identification and screening procedures outlined in this protocol. | From the invitation date until the end of the study (approximately 12 months).
  The primary objective of this study is to pilot the identification and screening procedures outlined in this protocol. This includes assessing the identification rate (%) and estimating the prevalence of heart failure with preserved ejection fraction (HFpEF) both overall and within different subgroups (%).

SECONDARY OUTCOMES:
Secondarily, we aim to assess the willingness of identified Danish adults with risk factors for HFpEF to participate in the study, as well as to identify and address any barriers to their involvement. | From the end of the study until all analyses are completed (estimated to be from November 2025 to March 2026
  * To assess response, acceptance, and attendance rates among participants, reported as percentages.
  * To investigate barriers to participation, categorizing and presenting them as percentages.
  * To analyze patterns among non-responders, using educational attainment, household income, and geographic distances to the study site as indicators of socioeconomic and sociodemographic status. All parameters will be clustered and reported as percentages.
  Through these objectives, we aim to gain a comprehensive understanding of participant engagement and identify any factors that may hinder participation in the screening process.

CONTACTS AND LOCATIONS:
Locations (1):
- Center for Translational Cardiology and Pragmatic Randomized Trials, Department of Cardiology, Copenhagen University Hospital, Herlev and Gentofte Hospital, Hellerup, Denmark

IPD SHARING:
Plan to Share IPD: Yes
Most data will be collected from Danish administrative health registries, which are subject to Danish legislation and can only be made available to a third party under certain conditions. Please contact the sponsor-investigator in case of any inquiries.